CLINICAL TRIAL: NCT07384104
Title: A Randomized, Open-Label, Single-Dose, Parallel-Controlled Biosimilarity Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of SAL023 and Italy-Manufactured Evenity in Healthy Adult Chinese Subjects
Brief Title: Compare the Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of SAL023 and Italy-Manufactured Evenity in Healthy Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Salubris (Chengdu) Biotechnology Co., Ltd. (Unknown); Salubris (Suzhou) Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAL023A102
Record Dates: First submitted 2026-01-13; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; Immunogenicity; Biosimilarity Comparison
MeSH Terms: conditions — Osteoporosis | interventions — romosozumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Drug: SAL0123 105mg:1.17ml
  Interventions: Drug: SAL0123
- Reference Group (Active Comparator): Drug: Romosozumab 105mg:1.17ml
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: SAL0123 — Dosage Form: Injection Specification: 105mg:1.17ml Dosage and Administration: 2 vials of 105 mg: 1.17 mL each, subcutaneous injection in the upper arm and abdomen Treatment Duration: Single subcutaneous injection of 2 vials on Day 1
  Arms: Test Group
Drug: Romosozumab — Dosage Form: Injection Specification: 105mg:1.17ml Dosage and Administration: 2 vials of 105 mg: 1.17 mL each, subcutaneous injection in the upper arm and abdomen Treatment Duration: Single subcutaneous injection of 2 vials on Day 1
  Arms: Reference Group

SUMMARY:
Primary objective of this study is to evaluate the similarity in pharmacokinetic characteristics between SAL023 Injection and Italy-manufactured Evenity. Secondary objective is to assess the similarity in safety, pharmacodynamic and immunogenicity profiles of SAL023 Injection and Italy-manufactured Evenity.

DETAILED DESCRIPTION:
This study adopts a randomized, open-label, single-dose, active-controlled, two-arm, parallel-group design.

The entire study will last approximately 16 weeks, consisting of a screening period, a dosing and inpatient observation period, and a follow-up period. A total of 118 healthy adult Chinese subjects are planned to be enrolled in the study and will be randomly assigned to the SAL023 group (Group A) and the Italy-manufactured Evenity group (Group B) at a ratio of 1:1, with 59 subjects in each group. All subjects will receive a single subcutaneous injection of either SAL023 or Italy-manufactured Evenity.

Eligible subjects will be admitted to the research center on Day -1 and undergo randomization. They will receive the required examinations on Day 10 after dosing, and will be discharged from the research center only after the investigator confirms their safety. After discharge, the subjects will return to the research center for regular follow-up visits in accordance with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of the study, voluntarily sign the written informed consent form (ICF), and be able to comply with the requirements and restrictions specified in the ICF.
2. Healthy Chinese male or female subjects.
3. Aged 18 to 45 years old (inclusive of both endpoints).
4. Body weight ≥ 50 kg and body mass index (BMI) ranging from 19.0 to 25.0 kg/m² (inclusive of both endpoints; BMI = weight ÷ height²).
5. Results of all examinations (including physical examination, vital signs, blood routine, urine routine, blood biochemistry, coagulation function, myocardial enzymes, thyroid function, serum virology, 12-lead electrocardiogram, chest X-ray (anteroposterior view), abdominal ultrasound, etc.) are normal or have minor abnormalities that are judged as not clinically insignificant by the investigator.
6. The subject or their partner has no pregnancy plans during the study period and within 3 months after the last administration of the study drug, and voluntarily adopts effective contraceptive measures (contraceptives are prohibited during the study period) to avoid pregnancy of themselves or their partner; in addition, the subject will not donate sperm or ova (egg cells, oocytes) for reproductive or assisted reproductive purposes.

Exclusion Criteria:

1. A history of clinically significant acute drug or food allergic reactions within 2 weeks prior to screening; or allergic diathesis (e.g., allergy to two or more drugs, foods or pollen); or a history of allergic diseases (e.g., asthma, urticaria, eczematous dermatitis, etc.); or a possible or definite allergy to the study drug (including similar drugs or the control drug) and any of its excipients, hypersensitivity reactions, or clinically significant notable reactions as judged by the investigator.
2. Positive result for any of the following tests: hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus antibody, or treponema pallidum antibody.
3. Bone mineral density T-score ≤ -2.5 at any of the following sites: lumbar vertebrae L1-L4 (total), total hip joint, or femoral neck during the screening period.
4. Serum calcium, creatinine, free triiodothyronine (FT3), free thyroxine (FT4), thyroid stimulating hormone (TSH), or parathyroid hormone levels outside the normal reference range.
5. A history of any of the following diseases: history of hip fracture or fracture at any other site within 6 months prior to the first administration; history of myocardial infarction; history of cerebral infarction or ischemic stroke.
6. Use of any of the following foods, drugs or treatments prior to the first administration: estrogen/progesterone replacement therapy, calcitonin, parathyroid hormone and its analogs, vitamin D supplements > 1000 IU/day, glucocorticoids (inhaled or topical glucocorticoids used more than 2 weeks before screening are allowed), anabolic steroids, calcitriol and its analogs, thiazide diuretics within 6 months prior to the first administration; bisphosphonates, fluoride for the treatment of osteoporosis within 12 months prior to the first administration; denosumab or any cathepsin K inhibitor within 18 months prior to the first administration; prior use of Romosozumab (including Evenity and other biosimilars); any prescription drugs or Chinese herbal medicines within 4 weeks prior to the first administration; any over-the-counter drugs and food supplements (including vitamins, calcium supplements, health food products, etc.) within 2 weeks prior to the first administration.
7. Drug or substance abuse, alcoholism or heavy smoking: history of drug or substance abuse, or positive result in drug abuse screening at the time of screening; average weekly alcohol consumption > 14 units within 3 months prior to screening (1 unit ≈ 17.7 mL ethanol, i.e., 1 unit ≈ 360 mL beer with 5% alcohol content, or 45 mL Baijiu (liquor) with 40% alcohol content, or 150 mL wine with 12% alcohol content), or positive alcohol test result at screening, or inability to completely abstain from any food or beverage containing alcohol during the hospitalization period; average daily cigarette consumption > 5 sticks within 3 months prior to screening, or inability to completely abstain from any tobacco products during the hospitalization period; average daily caffeine intake > 500 mg within 3 months prior to screening (equivalent to 5 cups of tea or coffee, or 8 cans of soda or other caffeinated products).
8. Blood donation (including component blood donation) or blood loss ≥ 400 mL within 3 months prior to screening; blood donation (including component blood donation) or blood loss ≥ 200 mL or blood transfusion within 1 month prior to screening; or plan to donate blood or blood components during the study period or within 1 month after the end of the study.
9. Difficulty in blood collection or inability to tolerate multiple venipunctures; or a history of clinically significant needle phobia or hematophobia as judged by the investigator.
10. Vaccination with live vaccines, live attenuated vaccines or any vaccine containing live viral components within 3 months prior to screening; or plan to receive the above vaccines during the study period or within 1 month after the end of the study.
11. Severe trauma or major surgery requiring general anesthesia within 3 months prior to screening; or plan to undergo surgery (except for surgery under local anesthesia) within 3 months after the last administration.
12. Participation in any interventional clinical study (including investigational drugs or vaccines, as well as other clinical studies of the study drug or other cohorts of this study) and receipt of investigational drugs within 3 months prior to screening, or current participation in such studies.
13. Other diseases or medical histories that are clinically significant or may prevent the subject from completing the study, or other diseases or medical histories that may significantly alter drug absorption, metabolism or excretion, as judged by the investigator.
14. Any other reasons that make the subject unsuitable for participation in this study, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-10-19 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
PK parameters（ Cmax） | Within a single dosing period ( from pre-dose up to 85 days post-dose)
PK parameters（ AUCinf） | Within a single dosing period ( from pre-dose up to 85 days post-dose)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University Clinical Pharmacology Research Center, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No